CLINICAL TRIAL: NCT07239570
Title: A Biomarker-targeted Clinical Trial to Optimize Treatment for Patients With Chronic Kidney Disease: A Prospective, Randomized, Open-Label, Parallel-Group, Multicenter Study
Brief Title: A Biomarker-targeted Clinical Trial to Optimize Treatment for Patients With Chronic Kidney Disease
Acronym: CKD-bioMatch
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peter Rossing (Other)
Collaborators: University Medical Center Groningen (Other); Lund University (Other); Instituto de Investigacion Sanitaria INCLIVA (Other); Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor-Investigator, Peter Rossing, Professor, MD, DMSc, Steno Diabetes Center Copenhagen
Organization: Steno Diabetes Center Copenhagen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-507449-27
Record Dates: First submitted 2025-04-30; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: Chronic Kidney Disease; Personalized medicine; Biomarkers
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — dapagliflozin; semaglutide; finerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Participants in the standard of care group will receive treatment following the KDIGO (Kidney Disease: Improving Global Outcomes) guidelines.
- Biomarker-targeted treatment (Experimental): In the treatment arm, the participants will receive stepwise treatment with one or more study drugs.
  The choice, order, and number of treatments introduced will be based on the participant's characteristics/risk profile and the response on UACR and UEGF.
  Interventions: Drug: Dapagliflozin; Drug: Semaglutide; Drug: Finerenone

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin 10 mg daily.
  Arms: Biomarker-targeted treatment
Drug: Semaglutide — Semaglutide injection once weekly. Will be titrated every 4 weeks to the highest tolerable dose according to standard guidelines, aiming at 1 mg once weekly.
  Arms: Biomarker-targeted treatment
Drug: Finerenone — Finerenone 10-20 mg daily.
  Arms: Biomarker-targeted treatment

SUMMARY:
Over 800 million people worldwide suffer from chronic kidney disease (CKD), which is associated with a high individual disease burden for those affected, multiple secondary diseases, frequent doctor contacts, and hospitalizations, but also outstanding costs for the health system and the solidarity community. Appropriate interventions are essential to prevent the development and progression of CKD. In the past decade, great progress has been made in the search for drugs that can slow the progression of CKD. Sodium-glucose co-transporter 2 inhibitors, the non-steroidal mineralocorticoid receptor antagonist, finerenone, and the glucagon-like peptide-1 receptor agonist, semaglutide, have demonstrated albuminuria-lowering effects and kidney protection in people with CKD. Although these new pharmacological approaches show great promise, it is unclear how to optimally sequence and combine these therapies. In addition, the therapies are often not implemented due to treatment inertia and fear of adverse effects. This study aims to address this knowledge gap by utilizing a biomarker-guided treatment approach to reduce the decline in kidney function.

The aim of the CKD-bioMatch study is to evaluate the efficacy of a biomarker-targeted treatment approach versus standard of care in people with CKD and albuminuria. We hypothesize that a biomarker-targeted treatment approach is superior to standard of care at reducing estimated glomerular filtration rate (eGFR) decline in people with CKD.

DETAILED DESCRIPTION:
The study is a prospective, randomized, open-label, parallel-group, multicenter study. CKD-bioMatch will enroll 125 individuals with CKD (eGFR ≥ 25 mL/min/1.73m² and UACR 100-5000 mg/g). Participants will be randomized 1:1 to a biomarker-targeted treatment approach versus standard of care.

In the treatment arm, a sequence of pharmacological treatments will be added (dapagliflozin, finerenone, and/or semaglutide), guided by the participant's characteristics and the urinary biomarkers urinary albumin-to-creatinine ratio (UACR) and urinary epidermal growth factor (UEGF). Participants will start treatment with one of the three study medications. After approximately four weeks on the maximum tolerated dose of the allocated medication, UACR and UEGF will be measured, and based on the biomarker response, a decision will be made to continue, switch, or add a new treatment. If a second drug is initiated, the treatment effect of that second drug will be evaluated on UACR and UEGF after four weeks on the maximum tolerated dose, and if the UACR response is insufficient, a third drug can be added, or the third drug can replace the second drug. The biomarker response of the third drug will be evaluated in the same manner as that of the first two drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 75 years
2. UACR 100-5000 mg/g (11.3-565 mg/mmol) in two consecutive first-morning void urine samples at screening. (UACR 80-100 mg/g is accepted if historical measurements are above 100 mg/g and if it cannot be explained by any new treatment.)
3. Stable treatment with a maximum tolerated dose of an angiotensin-converting enzyme inhibitor or angiotensin receptor blocker for at least four weeks prior to randomization. (Unless such treatment is contraindicated or not tolerated.)
4. Ability to communicate with the study staff and understand and sign the informed consent.

Exclusion Criteria:

1. eGFR < 25 mL/min/1.73m2 at screening.
2. Treatment with two or all three of the study drugs
3. History of pancreatitis at screening
4. Body mass index < 18.5 kg/m2 at screening
5. Type 1 diabetes
6. Myocardial infarction, unstable angina, stroke, or transient ischemic attack within 12 weeks prior to enrollment
7. NYHA class IV Congestive Heart Failure at screening
8. Potassium > 5.0 mmol/L at screening
9. Addison's Disease
10. Concomitant treatment with strong CYP3A4 inhibitors (e.g., itraconazole, ketoconazole, ritonavir, cobicistat, clarithromycin)
11. Treatment with a potassium-sparing diuretic or a mineralocorticoid receptor antagonist, except for finerenone (e.g., spironolactone, eplerenone, or amiloride)
12. Elevated Alanine Aminotransferase (ALT) > 3 x upper normal limit at screening, autoimmune hepatitis, and/or severe hepatic impairment (including but not limited to a history of hepatic encephalopathy, a history of esophageal varices, or a history of portocaval shunt).
13. Autosomal dominant or autosomal recessive polycystic kidney disease
14. Lupus nephritis or ANCA-associated vasculitis, or any other primary or secondary kidney disease requiring immunosuppressive therapy within 6 months prior to screening
15. Kidney transplant or dialysis
16. Known or suspected hypersensitivity to the study medications or related products
17. Presence or history of malignant neoplasms (except basal cell skin cancer or squamous cell skin cancer) within five years before screening.
18. Any other history, condition, therapy, or uncontrolled intercurrent illness that could, as judged by the investigator, affect participant safety or compliance with study requirements.
19. A female who is pregnant, breastfeeding, or intends to become pregnant, or a woman of childbearing potential (WOCBP) who is not using highly effective contraceptive methods.
20. Known or suspected abuse of narcotics.
21. Participant in another intervention study.
22. Vulnerable (i.e., under guardianship) or mentally incapacitated subjects (i.e., not able to understand and sign the informed consent).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Chronic eGFR slope | From week 26 to 104
  Mean annual rate of change in eGFR from week 26 to week 104.

SECONDARY OUTCOMES:
Change in eGFR from baseline to end of study | From baseline to week 112
  Change in eGFR from baseline to week 112 (end of study).
Change in eGFR from baseline to end of treatment. | From baseline to week 104
  Change in eGFR from baseline to week 104 (end of treatment).
Change in UACR | From baseline to week 104
  Change in UACR from baseline to week 104 (end of treatment)

OTHER OUTCOMES:
Change in KidneyIntelX score | From baseline to week 104
  Change in KidneyIntelX (kidney risk score) score from baseline to week 104 (end of treatment). An increase in the score represents an increase in predicted risk of CKD progression, and a decline represents a reduction in predicted risk.

CONTACTS AND LOCATIONS:
Locations (4):
- Steno Diabetes Center Copenhagen, Herlev, Denmark
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany
- Hospital Clinico de Valencia, Valencia, Spain
- Lund University, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://prime-ckd.com/